CLINICAL TRIAL: NCT00205192
Title: Optimizing Cardiac Resynchronization
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2004-0335
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiac resynchronization; echocardiography
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cardiac resynchronization pacing — various pacemaker modes used over 1 hour

SUMMARY:
Cardiac resynchronization therapy shows great promise as a method to improve ventricular function in heart failure due to dilated cardiomyopathy. It is applied to patients with class III and IV symptomatic heart failure on optimal therapy. Typical entry criteria in the trials testing resynchronization have used the electrocardiogram and a prolonged electrocardiogram (ECG) QRS interval as criteria for dyssynchrony. This is recognized to be quite limited as a tool for identifying patients. Several new echocardiographic methods for identifying dyssynchrony have been proposed. The purpose of this study is to systematically examine these multiple echocardiographic measurement techniques in three conditions:

1. in the patient's native rhythm simulated by changing the pacing system to atrial pacing only;
2. in conventional dual chamber pacing (DDD mode); and
3. during biventricular pacing. All patients entered into this study will already have had a biventricular pacemaker placed.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have previously had a resynchronization pacemaker system placed at the University of Wisconsin Hospital or at the Middleton Veterans Hospital are potentially eligible for this study.
* The study is only open to patients as enumerated above, and also patients who have good imaging windows.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have previously had a resynchronization pacemaker system placed at the University of Wisconsin Hospital or at the Middleton Veterans Hospital are potentially eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2004-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Rahko, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States